CLINICAL TRIAL: NCT01725503
Title: Creatine Metabolism in Humans:Effect of Creatine and Amino Acid Supplement
Brief Title: Creatine Kinetics, Synthesis From Glycine and Response to Creatine and Amino Acid Supplement in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Satish Kalhan, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-005
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Creatine Synthesis in Healthy Subjects
Keywords: creatine synthesis
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Creatine and amino acid supplement (Experimental)
  Interventions: Dietary Supplement: Creatine and Amino Acid supplement

INTERVENTIONS:
Dietary Supplement: Creatine and Amino Acid supplement

SUMMARY:
The goal of the present study is to quantify the rate of synthesis of creatine in healthy controls and endurance trained subjects. In addition, the effect of oral creatine supplement for seven days on creatine kinetics will be examined.

Ten healthy controls (age 20-35 years) and ten endurance trained subjects will be recruited by advertisement. Endurance trained subjects will be recruited from health clubs. They will be screened for absence of any chronic disease (history, physical examination, CBC, metabolic and liver panel, urinalysis). A DEXA measurement will be done to quantify whole body skeletal muscle mass.

For five (5) days prior to the study, they will be placed on a creatine-free (essentially meat-free) diet. Dietary compliance will be ensured by repeated communication with the subject, by nurse coordinator and the CRU Nutritionist. Subject will maintain daily record of the food intake for validation. On the last day, i.e. 24 hours prior to the tracer study, subject will collect the 24 hours urine sample and bring it to the CRU on the day of the study.

DETAILED DESCRIPTION:
Creatine and phosphocreatine are the major intracellular buffers for adenosine triphosphate. They also function as the energy shuttle for high energy phosphate from the mitochondrial site of production to the cytoplasmic site of utilization. In addition, creatine has been shown to affect satellite cell proliferation and differentiation and increase cell mitotic activity during compensatory hypertrophy in rat skeletal muscle. Creatine is synthesized from three amino acids: glycine, arginine and methionine. Although creatine metabolism has been studied extensively in the rat, the data regarding the kinetics of creatine and their regulation in humans are limited. This is in part due to a large and slow turning over pool of creatine and lack of good tracer methods. Using a recently developed stable isotopic tracer method (by us), we propose to quantify the rate of synthesis of creatine and its regulation in healthy subjects and in those with large skeletal muscle mass as a result of endurance training. In addition, the response to oral creatine administration on creatine kinetics will be quantified. The site of regulation will be identified by the relative rate of appearance of tracer glycine in guanidinoacetic acid and creatine. It is hypothesized that the fractional rate of synthesis of creatine will be higher in endurance trained subjects, and that creatine will suppress the rate of synthesis of creatine. Since creatine is critical for the maintenance of skeletal muscle mass and satellite cell proliferation, these data will provide the normative physiological data for future studies of subjects with manifest sarcopenia, such as aging, and those with chronic diseases, e.g. cirrhosis of liver. These data will form the basis for the studies of creatine metabolism in neurodegenerative disorders where creatine is being increasingly used as a therapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls and endurance trained subjects
* Both males and females will be studied.

Exclusion Criteria:

* any illness
* on any medications and/or supplements

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quantification of creatine synthesis in healthy subjects | 12/31/2012

SECONDARY OUTCOMES:
Effect of creatine supplement on the rate of creatine synthesis | 12/31/2012

CONTACTS AND LOCATIONS:
Overall Officials: Satish Kalhan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States